CLINICAL TRIAL: NCT03403777
Title: Phase II Study of Avelumab in Multiple Relapsed/Refractory Testicular Germ Cell Cancer.
Brief Title: Avelumab in Refractory Testicular Germ Cell Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCISlovakia
Record Dates: First submitted 2018-01-02; First posted 2018-01-19 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal; Neoplasms; Testicular Diseases; Gonadal Disorders; Antineoplastic Agents; Molecular Mechanisms of Pharmacological Action
Keywords: Multiple relapsed/refractory testicular germ cell tumors; Avelumab; Anti PD-L1
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal; Neoplasms; Testicular Diseases; Gonadal Disorders | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Non-randomized, open-label, multi-centre trial to assess efficacy (as measured by 12-week progression-free survival) of AVELUMAB in patients with refractory germ cell tumors (GCTs). The Simon optimal 2-stage design (see statistical section) will be used. See section 6 (Statistical Considerations) for specific details.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab (Experimental): AVELUMAB will be administered intravenously 10mg/kg every 2 weeks. Courses will be repeated every 14 days until progression or unacceptable toxicity. AVELUMAB will be administered as a 1-hour (-10 minutes / +20 minutes, i.e., 50-80 minutes) intravenous (i.v.) infusion. The dose of AVELUMAB will be calculated based on the weight of the subject determined on the day prior to or the day of each drug administration.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — AVELUMAB will be administered intravenously 10mg/kg every 2 weeks.
  Other Names: Bavencio

SUMMARY:
This is a proof-of-concept study to define efficacy of AVELUMAB in patients with multiple relapsed/refractory germ cell tumors (GCTs). Data suggest that PD-L1 is overexpressed in TGCTs, and PD-L1 expression is significantly higher in GCTs in comparison to normal testicular tissue.Patients with low PD-L1 expression had significantly better progression-free survival (hazard ratio [HR] = 0.40, 95% CI (0.16 - 1.01, p = 0.008) and overall survival (HR = 0.43, 95% CI (0.15 - 1.23, p = 0.040) compared to patients with high PD-L1 expression. These data suggest that PD-1/PD-L1 pathway could be a novel therapeutic target in TGCTs and that there is strong rationale to inhibit PD-1/PD-L1 signaling in GCTs.

DETAILED DESCRIPTION:
Germ-cell tumours (GCTs) are extraordinarily chemosensitive and resemble the clinical and biological characteristics of a model for the cure of cancer. Nonetheless, a small proportion of patients do not have a durable complete remission (CR) with initial chemotherapy. Only 20-40% of them will be cured with the use of platinum-containing standard-dose or high-dose salvage chemotherapy with autologous stem cell transplantation (ASCT). Patients who fail to be cured after second-line salvage therapy have an extremely poor prognosis and long term survival had been documented in <5%. Paclitaxel plus ifosfamide and cisplatin is considered as a standard salvage chemotherapy in relapsed good prognosis GCTs, however, up to 40% of favourable prognosis patients failed to achieve durable response to this combination, and therefore new treatment strategies are warranted.

Recent data suggest that PD-L1 is overexpressed in TGCTs, including 73% seminomas and 64% non-seminomatous tumors, but none of normal testicular tissue specimens exhibited PD-L1 expression. In previous study that included 140 patients, PD-L1 was significantly higher in GCTs in comparison to normal testicular tissue (mean QS = 5.29 vs. 0.32, p < 0.0001). Choriocarcinomas exhibit the highest level of PD-L1 with decreasing positivity in embryonal carcinoma, teratoma, yolk sac tumor and seminoma. PD-L1 expression was associated with poor prognostic features including ≥ 3 metastatic sites, increased serum tumor markers and/or non-pulmonary visceral metastases. Patients with low PD-L1 expression had significantly better progression-free survival (hazard ratio [HR] = 0.40, 95% CI (0.16 - 1.01, p = 0.008) and overall survival (HR = 0.43, 95% CI (0.15 - 1.23, p = 0.040) compared to patients with high PD-L1 expression (Figure 1).

These data suggest that PD-1/PD-L1 pathway could be a novel therapeutic target in TGCTs and that there is strong rationale to inhibit PD-1/PD-L1 signaling in GCTs and phase II study is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Men aged 18 years or older
3. ECOG performance status: 0-1
4. Histologically confirmed extracranial primary germ cell cancer, seminoma, or nonseminoma
5. Rising serum markers (i.e., alpha-fetoprotein and human chorionic gonadotropin) on sequential measurement or biopsy-proven unresectable germ cell cancer
6. Refractory GCTs e.g. patients relapsing after high-dose chemotherapy or for patients non fit enough for high-dose chemotherapy
7. Primary mediastinal GCTs in first relapse
8. Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of investigator,
9. RECIST 1.1 Measurable disease
10. Adequate hematologic function defined by ANC ≥ 1500/mm3, platelet count ≥ 100 000/mm3 and hemoglobin level ≥ 9g/dl.
11. Adequate liver function defined by a total bilirubin level ≤ 1.5 ULN, and ALT, AST ≤ 2.5 × ULN . or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
12. Adequate renal function: measured or calculated (by Cockcroft formula) creatinine clearance ≥ 30 ml/min. Cockcroft formula: CLcr = [(140-age) x weight(Kg)]/[72 x creat (mg/dl)]
13. At least 4 weeks must have elapsed since the last radiotherapy and/or chemotherapy before study entry,
14. At least 4 weeks must have elapsed since the last major surgery
15. Complete recovery from prior surgery, and/or reduction of all adverse events from previous systemic therapy or radiotherapy to grade 1,
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
17. Highly effective contraception for both male and female subjects if the risk of conception exists. (Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraception, defined as methods with a failure rate of less than 1 % per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 30 days after avelumab treatment.

Exclusion Criteria:

1. Patients who do not fit inclusion criteria
2. Other prior malignancy except successfully treated non-melanoma skin cancer
3. No prior PD-1/PD-L1 inhibitor
4. Other concurrent approved or investigational anticancer treatment, including surgery, radiotherapy, chemotherapy, biologic-response modifiers, hormone therapy, or immunotherapy
5. Female patients
6. Patients infected by the Human Immunodeficiency Virus (HIV)
7. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
8. Other significant diseases: e.g. immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; Patients with other severe acute or chronic medical condition, or laboratory abnormality that would impair, in the judgment of investigator, excess risk associated with the study participation, study treatment administration, or may interfere with the interpretation of study results and, which, in judgment of the investigator, would make the patient inappropriate for entry into this study.
9. Hypersensitivity to any compound of the drug
10. Sexually active men not using highly effective birth control if their partners are women of child-bearing potential
11. All subjects with brain metastases, except those meeting the following criteria:

    * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
    * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
    * Subjects must be either off steroids or on a stable or decreasing dose of <10mg daily prednisone (or equivalent)
12. Prior organ transplantation, including allogeneic stem cell transplantation
13. Significant acute or chronic infections including, among others:
14. Active infection requiring systemic therapy

    * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
    * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
15. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

    1. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
    2. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
    3. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation...) are acceptable
    4. steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
16. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
17. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable
18. Known alcohol or drug abuse
19. All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment
20. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
21. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy (as measured by 12-week progression-free survival) of AVELUMAB in patients with multiple relapsed/refractory germ cell tumors (GCTs). | 12-weeks
  12-week progression-free survival

SECONDARY OUTCOMES:
To describe the favorable response rate of AVELUMAB in patients with multiple relapsed/refractory germ cell tumors (GCTs). | 4-weeks
  Favorable response rate - complete remission and/or partial remission with negative serum tumor markers
Progression-free survival (PFS) of AVELUMAB in patients with multiple relapsed/refractory germ cell tumors (GCTs). | 12-months
  Progression-free survival (PFS) will be calculated from the beginning of the treatment until progression or death from disease-specific cause on intention-to-treat basis.
Toxic effects of AVELUMAB in patients with multiple relapsed/refractory germ cell tumors (GCTs). | 12-weeks
  Toxicity according to NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, prof, Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) Broun ER et al. Ann Intern Med 1993; 117: 124-8 2) Cierna et al., Ann Oncol, Ann Oncol. 2016 Feb;27(2):300-5. 3) Feldman et al Cancer 2012;118:981-6. 4) Horwich A, et al. Lancet 2006; 367: 754-65 5) Kollmannsberger C et al. Cancer 2006; 106: 1217-26 6) Kondagunta GV et al. J Clin Oncol. 2005 23:6549-55. 7) Mardiak J et al. Neoplasma, 2005; 52: 497-501 8) Fankhauser, C. D et al. Br J Cancer. 2015, 113: 411-413 9) Heery et al. J Clin Oncol 33, 2015 (suppl; abstr 3055) 10) Yamada et al. J Clin Oncol 33, 2015 (suppl; abstr 4047) 11) Disis et al. J Clin Oncol 33, 2015 (suppl; abstr 5509) 12) Gulley et al. J Clin Oncol 33, 2015 (suppl; abstr 8034) 13) Shitara K et al. J Clin Oncol 33, 2015 (suppl; abstr 3023) 14) Kelly K et al. J Clin Oncol 33, 2015 (suppl; abstr 3044) 15) Boyerinas B et al. Cancer Immunol Res. 2015 Oct;3(10):1148-57.